CLINICAL TRIAL: NCT06025695
Title: A Phase III, Observer-blind, Randomized, Multicenter Study to Evaluate Immunogenicity, Reactogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Rotarix Porcine Circovirus (PCV)-Free Liquid as Compared to GSK's Rotarix Liquid, Given in 2-doses in Healthy Chinese Infants Starting at Age 6-16 Weeks
Brief Title: Immunogenicity, Reactogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Rotarix Porcine Circovirus (PCV)-Free Liquid Compared to Rotarix Liquid Given in 2-doses in Healthy Chinese Infants Starting at Age 6-16 Weeks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 212692; 2020-000972-38 (EudraCT Number)
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Gastroenteritis
Keywords: Rotavirus (RV); Human rotavirus (HRV); Rotarix Porcine circovirus (PCV)-free liquid; Rotarix liquid; Healthy Chinese infants; Immunogenicity; Reactogenicity; Safety
MeSH Terms: conditions — Gastroenteritis | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be conducted in an observer-blind manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Human Rotavirus (HRV) Group (Active Comparator): Participants received 2 doses of GSK's liquid oral live attenuated HRV study intervention at Day 1 and Month 1.
  Interventions: Combination Product: GSK's liquid oral live attenuated HRV
- HRV Porcine Circovirus (PCV)-free Group (Experimental): Participants received 2 doses of the PCV-free liquid formulation of GSK's oral live attenuated HRV study intervention at Day 1 and Month 1.
  Interventions: Combination Product: PCV-free liquid formulation of GSK's oral live attenuated HRV

INTERVENTIONS:
Combination Product: GSK's liquid oral live attenuated HRV — 2 doses of GSK's liquid oral live attenuated HRV study intervention administered orally at Day 1 and Month 1, according to the immunization schedule for HRV study intervention licensed outside of China.
  Other Names: Rotarix
  Arms: Human Rotavirus (HRV) Group
Combination Product: PCV-free liquid formulation of GSK's oral live attenuated HRV — 2 doses of PCV-free liquid formulation of GSK's oral live attenuated HRV study intervention administered orally at Day 1 and Month 1, according to the immunization schedule for HRV study intervention licensed outside of China.
  Other Names: Rotarix PCV-free
  Arms: HRV Porcine Circovirus (PCV)-free Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, reactogenicity and safety of the Porcine circovirus (PCV)-free liquid formulation of GlaxoSmithKline Biologicals' SA (GSK) oral live attenuated human rotavirus (HRV) study intervention compared to GSK's liquid oral live attenuated HRV study intervention in healthy Chinese infants 6 to 16 weeks of age at the time of the first study intervention administration.

ELIGIBILITY:
Inclusion Criteria:

* Participants' parent(s)/legally acceptable representative(s) [LAR(s)], who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the parent(s)/LAR(s) of the participant prior to performance of any study specific procedure.
* A male or female with Chinese origin, between, and including, 6 and 16 weeks (42-112 days) of age at the time of the first study intervention administration.
* Healthy participants as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of 36 to 42 weeks inclusive.

Exclusion Criteria:

Medical conditions

* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of severe combined immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention.
* History of seizures or progressive neurological disease.
* Family history of congenital or hereditary immunodeficiency.
* Uncorrected congenital malformation of the gastrointestinal tract that would predispose for intussusception (IS).
* History of IS.
* Major congenital defects, or serious chronic illness as assessed by the investigator.
* Previous confirmed occurrence of rotavirus gastroenteritis (RVGE).
* Participants with confirmed or suspected Coronavirus Disease 2019 (COVID-19).

Prior/Concomitant therapy

* Use of any investigational or non-registered product other than the study interventions during the period beginning 30 days before the first dose of study interventions (Day -29 to Day 1), or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the second dose of study intervention administration*, with the exception of the inactivated influenza vaccine, which is allowed at any time during the study and other licensed routine childhood vaccinations.

  *In case emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is organized by public health authorities outside the routine immunization programme, the time period described above can be reduced if, necessary for that mass vaccination vaccine, provided it is licensed and used according to its Product Information.
* Administration of immunoglobulins and/or any blood products or plasma derivatives from birth or planned administration during the study period.
* Administration of long-acting immune-modifying drugs from birth or planned administration at any time during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth. For corticosteroids, this will mean prednisone >= 0.5 milligram/kilogram (kg)/day, or equivalent. Inhaled and topical steroids are allowed.
* Previous vaccination against RV.

Prior/Concurrent clinical study experience

- Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product.

Other exclusions

- Child in care.

Ages: 6 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - GSK Investigational Site, Baoshan
  - GSK Investigational Site, Dali
  - GSK Investigational Site, Honghe
  - GSK Investigational Site, Mianyang
  - GSK Investigational Site, Nanbu-Nanchong
  - GSK Investigational Site, Neijiang
  - GSK Investigational Site, Tengchong
  - GSK Investigational Site, Wenshan

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in China.
Pre-assignment Details: One participant was randomized to the HRV group but was vaccinated in the HRV PCV-free group. Data for this participant was analyzed in the HRV PCV-free group for all analyses.
Period: Overall Study
Arm/Group | Human Rotavirus (HRV) Group | HRV Porcine Circovirus (PCV)-Free Group
Started | 998 | 1002
Completed | 956 | 967
Not Completed | 42 | 35
Not completed — Adverse Event | 5 | 6
Not completed — Migrated / Moved from the Study Area | 13 | 10
Not completed — Other | 23 | 19
Not completed — Adverse Event Requiring Expedited Report | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Human Rotavirus (HRV) Group | HRV Porcine Circovirus (PCV)-Free Group | Total
Number analyzed (Participants) | 998 | 1002 | 2000
Age, Continuous [Mean (Standard Deviation); unit: WEEKS] | 10.1 (2.9) | 10.2 (2.9) | 10.1 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 455 | 512 | 967
  Male | 543 | 490 | 1033
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN - EAST ASIAN HERITAGE | 998 | 1002 | 2000

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Anti-rotavirus (RV) Immunoglobulin A (IgA) Antibody (Ab) Seroconversion Rate
Description: Seroconversion rate is defined as the percentage of participants who were initially seronegative (i.e., with anti-RV IgA Ab concentration below [<] 20 unit per milliliter [U/mL] prior the first dose of study intervention) and developed anti-RV IgA Ab concentration greater than or equal to (>=) 20 U/mL at Month 2 (1-month post-Dose 2).
Time Frame: At Month 2 (1-month post-Dose 2)
Population: Analysis was performed on Per Protocol Set (PPS), which includes all participants who adhered to the study protocol, ensuring they received no unapproved treatments, remained blinded, had anti-RV concentration <20 U/mL before intervention, had available anti-RV results at Month 2, complied with blood sampling schedules, and had no concurrent infections. Only participants with data available at specified timepoints were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Human Rotavirus (HRV) Group | HRV Porcine Circovirus (PCV)-Free Group
Number analyzed (Participants) | 865 | 870
Percentage of participants | 88.7 [86.4 to 90.7] | 84.9 [82.4 to 87.3]
Statistical Analysis 1: Comparison: Human Rotavirus (HRV) Group vs HRV Porcine Circovirus (PCV)-Free Group; To demonstrate the immunological non-inferiority of HRV PCV-free Group as compared to HRV Group in terms of seroconversion rates 1 month post-Dose 2; Test type: Non-Inferiority — Non-inferiority (NI) was to be demonstrated if the lower limit (LL) of the two-sided asymptotic standardized 95% confidence interval (CI) for the difference in seroconversion rate between the HRV PCV-free group and HRV group is greater than or equal to -10%; Difference in seroconversion rate = -3.73, 95% CI 2-sided [-6.93 to -0.55] — The asymptotic standardized 95% CI for the difference in seroconversion rate between HRV PCV-free Group minus HRV Group is computed using the method of Miettinen and Nurminen

2. Primary Outcome: Serum Anti-RV IgA Ab Concentrations Expressed as Geometric Mean Concentrations (GMCs)
Time Frame: At Month 2 (1-month post-Dose 2)
Population: Analysis was performed on PPS. Only participants with data available at the specified timepoints were included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Human Rotavirus (HRV) Group | HRV Porcine Circovirus (PCV)-Free Group
Number analyzed (Participants) | 865 | 870
U/mL | 222.82 [198.03 to 250.71] | 157.31 [139.31 to 177.64]
Statistical Analysis 1: Comparison: Human Rotavirus (HRV) Group vs HRV Porcine Circovirus (PCV)-Free Group; To demonstrate the non-inferiority of the HRV PCV-free Group as compared to HRV Group in terms of serum anti-RV IgA Ab concentrations 1 month post-Dose 2; Test type: Non-Inferiority — NI was to be demonstrated if the LL of the two-sided 95% CI for the ratio of anti-RV IgA Ab GMC between the HRV PCV-free group and HRV group is greater than or equal to 0.67; GMC Ratio = 0.71, 95% CI 2-sided [0.60 to 0.84] — The comparison is done using the group GMC ratio (HRV PCV-free/HRV) (ANOVA model applied to the log10-transformed titers). The ANOVA model included the group as a fixed effect

3. Secondary Outcome: Percentage of Participants With Serum Anti-RV IgA Ab Concentrations >= 90 U/mL
Time Frame: At Month 2 (1-month post-Dose 2)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Human Rotavirus (HRV) Group | HRV Porcine Circovirus (PCV)-Free Group
Number analyzed (Participants) | 865 | 870
Percentage of participants | 69.2 [66.1 to 72.3] | 62.9 [59.6 to 66.1]
Statistical Analysis 1: Comparison: Human Rotavirus (HRV) Group vs HRV Porcine Circovirus (PCV)-Free Group; To demonstrate the immunological non-inferiority of HRV PCV-free Group as compared to HRV Group in terms of percentage of participants with anti-RV IgA antibody concentrations >=90 U/mL 1 month post-Dose 2; Test type: Non-Inferiority — NI was to be demonstrated if the LL of the two-sided asymptotic standardized 95% CI for the difference in the percentage between the HRV PCV-free group and HRV group is greater than or equal to -10%; Difference in percentage = -6.37, 95% CI 2-sided [-10.81 to -1.92] — The asymptotic standardized 95% CI for the difference in in the percentage between HRV PCV-free Group minus HRV Group is computed using the method of Miettinen and Nurminen

4. Secondary Outcome: Number of Participants Reporting Solicited Systemic Events
Description: Solicited systemic events include fever/pyrexia, diarrhoea, vomiting, irritability/fussiness, loss of appetite, cough/runny nose. Fever is defined as body temperature >= 37.5 degrees Celsius (°C) and the preferred location for measuring temperature is the axilla. Any = occurrence of the event regardless of intensity grade or relation to the study vaccination.
Time Frame: Within 14 days (the day of vaccination and 13 subsequent days) after each vaccination (occurring at Day 1 and Month 1)
Population: Analysis was performed on the Exposed Set which includes all participants with at least 1 dose of the study intervention administered and with the solicited systemic events diary card data available after the corresponding vaccination for the specified timepoint. Only participants with data available at the specified timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Human Rotavirus (HRV) Group | HRV Porcine Circovirus (PCV)-Free Group
Number analyzed (Participants) | 973 | 986
Participants
  Cough/Runny Nose, post vaccination at Day 1 | 158 | 200
  Cough/Runny Nose, post vaccination at Month 1: number analyzed (Participants) | 956 | 961
  Cough/Runny Nose, post vaccination at Month 1 | 131 | 157
  Diarrhoea, post vaccination at Day 1 | 66 | 66
  Diarrhoea, post vaccination at Month 1: number analyzed (Participants) | 956 | 961
  Diarrhoea, post vaccination at Month 1 | 38 | 40
  Fever/Pyrexia, post vaccination at Day 1 | 122 | 100
  Fever/Pyrexia, post vaccination at Month 1: number analyzed (Participants) | 956 | 961
  Fever/Pyrexia, post vaccination at Month 1 | 104 | 91
  Irritability/Fussiness, post vaccination at Day 1 | 126 | 150
  Irritability/Fussiness, post vaccination at Month 1: number analyzed (Participants) | 956 | 961
  Irritability/Fussiness, post vaccination at Month 1 | 61 | 59
  Loss of appetite, post vaccination at Day 1 | 73 | 92
  Loss of appetite, post vaccination at Month 1: number analyzed (Participants) | 956 | 961
  Loss of appetite, post vaccination at Month 1 | 32 | 34
  Vomiting, post vaccination at Day 1 | 71 | 69
  Vomiting, post vaccination at Month 1: number analyzed (Participants) | 956 | 961
  Vomiting, post vaccination at Month 1 | 30 | 36

5. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AEs include any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event. Any = occurrence the event regardless of intensity grade or relation to the study vaccination
Time Frame: Within 31 days (the day of vaccination and 30 subsequent days) after each vaccination (occurring at Day 1 and Month 1)
Population: Analysis was performed on the Exposed Set which includes all participants with at least 1 dose of the study intervention administered and for whom unsolicited AEs data were available after the corresponding vaccination for the specified timepoint. Only participants with data available at the specified timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Human Rotavirus (HRV) Group | HRV Porcine Circovirus (PCV)-Free Group
Number analyzed (Participants) | 998 | 1002
Participants
  Post-vaccination at Day 1 | 236 | 234
  Post-vaccination at Month 1: number analyzed (Participants) | 965 | 970
  Post-vaccination at Month 1 | 223 | 229

6. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity or in other situations that are considered serious as per medical or scientific judgment. Any = occurrence of the SAE regardless of intensity grade or relation to the study vaccination.
Time Frame: From Day 1 to Month 7
Population: Analysis was performed on the Exposed Set which includes all participants with at least 1 dose of the study intervention administered and for whom SAE data were available after the corresponding vaccination for the specified timepoint. Only participants with data available at the specified timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Human Rotavirus (HRV) Group | HRV Porcine Circovirus (PCV)-Free Group
Number analyzed (Participants) | 998 | 1002
Participants | 251 | 262

ADVERSE EVENTS:
Time Frame: Solicited AEs: during the 14-day follow-up period (from Day 1 to Day 14) after any vaccination and unsolicited AEs: during the 31-day follow-up period after any vaccination (from Day 1 to Day 31). All cause mortality and SAEs were collected from Day 1 to Month 7.
Description: SAEs, solicited AEs and unsolicited AEs were reported for the Exposed set.
Arm/Group | Human Rotavirus (HRV) Group | HRV Porcine Circovirus (PCV)-Free Group
All-Cause Mortality (participants affected / at risk) | 1/998 | 0/1002
Serious Adverse Events (participants affected / at risk) | 251/998 | 262/1002
Other Adverse Events (participants affected / at risk) | 596/998 | 617/1002
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Rotavirus (HRV) Group (N=998) | HRV Porcine Circovirus (PCV)-Free Group (N=1002)
Pneumonia (Infections and infestations) | 140 (163) | 138 (160)
Bronchitis (Infections and infestations) | 39 (41) | 36 (37)
Febrile infection (Infections and infestations) | 21 (23) | 20 (22)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 11 (12)
Pharyngitis (Infections and infestations) | 5 (5) | 13 (14)
Gastroenteritis (Infections and infestations) | 6 (6) | 6 (6)
Pneumonia bacterial (Infections and infestations) | 6 (6) | 6 (6)
Gastrointestinal infection (Infections and infestations) | 3 (3) | 8 (8)
Laryngitis (Infections and infestations) | 7 (7) | 3 (3)
Herpangina (Infections and infestations) | 3 (3) | 5 (6)
Laryngopharyngitis (Infections and infestations) | 6 (6) | 1 (1)
Sepsis (Infections and infestations) | 5 (6) | 2 (2)
Gastroenteritis rotavirus (Infections and infestations) | 3 (3) | 4 (4)
Pneumonia haemophilus (Infections and infestations) | 3 (3) | 4 (4)
COVID-19 (Infections and infestations) | 2 (2) | 5 (5)
Influenza (Infections and infestations) | 1 (1) | 6 (6)
Respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3)
Enterobacter pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Pneumonia escherichia (Infections and infestations) | 4 (5) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 2 (2) | 2 (2)
Tracheobronchitis mycoplasmal (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia mycoplasmal (Infections and infestations) | 2 (2) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia respiratory syncytial viral (Infections and infestations) | 2 (2) | 0 (0)
Tracheitis (Infections and infestations) | 2 (2) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1)
Exanthema subitum (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Pertussis (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 2 (2)
Coxsackie viral infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Mycoplasma infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial diarrhoea (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia moraxella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 6 (6) | 5 (5)
Infantile diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7)
Cardiac failure (Cardiac disorders) | 1 (1) | 4 (4)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 2 (2) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Congenital megacolon (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Craniosynostosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vascular malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Rotavirus (HRV) Group (N=998) | HRV Porcine Circovirus (PCV)-Free Group (N=1002)
Respiratory tract infection (Infections and infestations) | 181 (203) | 219 (255)
Upper respiratory tract infection (Infections and infestations) | 46 (48) | 45 (55)
Bronchitis (Infections and infestations) | 13 (13) | 14 (14)
Pharyngitis (Infections and infestations) | 14 (15) | 9 (9)
Nasopharyngitis (Infections and infestations) | 8 (8) | 9 (9)
Gastroenteritis (Infections and infestations) | 8 (8) | 7 (7)
Laryngitis (Infections and infestations) | 4 (4) | 4 (4)
Pneumonia (Infections and infestations) | 2 (2) | 6 (6)
Candida infection (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 2 (2)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Dacryocystitis (Infections and infestations) | 1 (1) | 0 (0)
Dermatitis infected (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Eczema infected (Infections and infestations) | 1 (1) | 0 (0)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Herpangina (Infections and infestations) | 1 (1) | 0 (0)
Mycoplasma infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Chlamydial infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 123 (133) | 118 (131)
Vomiting (Gastrointestinal disorders) | 85 (98) | 95 (106)
Constipation (Gastrointestinal disorders) | 13 (13) | 18 (18)
Dyspepsia (Gastrointestinal disorders) | 9 (9) | 7 (7)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 3 (3)
Infantile diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 3 (4) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 3 (4)
Enteritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infantile colic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 91 (96) | 87 (94)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 61 (62) | 81 (86)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 35 (39) | 25 (26)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 13 (14)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 6 (8)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoventilation neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 178 (201) | 178 (195)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 149 (179) | 155 (191)
Sleep terror (Psychiatric disorders) | 0 (0) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 91 (104) | 102 (114)
Electrolyte imbalance (Metabolism and nutrition disorders) | 4 (5) | 8 (8)
Hyperlactacidaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Acid-base balance disorder mixed (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 17 (19) | 18 (18)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema infantile (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pityriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Myocardial necrosis marker increased (Investigations) | 10 (11) | 9 (9)
Immunoglobulins decreased (Investigations) | 2 (2) | 2 (2)
Liver function test abnormal (Investigations) | 1 (1) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 1 (1)
Bile acids increased (Investigations) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Secondary thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myocardial injury (Cardiac disorders) | 3 (3) | 7 (7)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 4 (4) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hypercholia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 3 (3) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Congenital laryngeal stridor (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Congenital laryngeal malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (2)
Transient hypogammaglobulinaemia of infancy (Immune system disorders) | 2 (2) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Drooling (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Transient neonatal hyperthyrotropinaemia (Endocrine disorders) | 1 (1) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT06025695/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT06025695/SAP_001.pdf